CLINICAL TRIAL: NCT01416597
Title: Effect of Influenza Vaccine Against Mismatched Strains: Systematic Review
Brief Title: A Systematic Review of Studies of the Effect of Influenza Vaccine Against Mismatched Strains
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115997
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Influenza
Keywords: Influenza; Systematic review; Meta-analysis; Mismatched strains; Cross-protection
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines

GROUPS / COHORTS (1):
- Cross-Protection Studies
  Interventions: Biological: Vaccines

INTERVENTIONS:
Biological: Vaccines — Unadjuvanted, monovalent, and trivalent vaccines, and vaccines delivered intramuscularly, intradermally, or intranasally, depending on what is found in the included studies.

SUMMARY:
The purpose of this study is to consolidate the cross-protection offered by influenza vaccines against circulating influenza A or B viruses that are not antigenically well-matched to vaccine strains and to determine the degree of cross-protection separately for influenza A and influenza B, through a systematic review of the literature.

DETAILED DESCRIPTION:
The research question of this project is: "what is the cross-protection afforded by vaccination (using an LAIV, TIV, or other type of vaccine) against influenza A or B and their subtypes and lineages?" The Preferred Reporting Items for Systematic Reviews and Meta-analyses (PRISMA) Statement will be used to guide the reporting of this review. Studies reporting cross-protection data after vaccination with approved formulations of influenza vaccines with influenza A or B will be included. Inclusion will not be limited by publication status, or year of dissemination but will be limited to randomized clinical trials (RCTs) and quasi-RCTs comparing influenza vaccine(s) with placebo. Only RCTs written in English will be included. A meta-analysis will be conducted if there is sufficient data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, adults or the elderly will be included that participated in randomized clinical trials (RCTs) and quasi-RCTs comparing influenza vaccine(s) with placebo.
* Placebo-controlled randomized clinical trials (RCTs) reporting laboratory-confirmed influenza among healthy participants vaccinated with antigens of influenza strains that differed from those circulating.
* All influenza vaccines will be included, and will be categorized as TIV, LAIV, and others (that is, non-TIV or non-LAIV).
* Only RCTs written in English will be included.

Exclusion Criteria:

* RCTs which are not providing any data will be excluded.
* Studies using rapid influenza diagnostic tests will not be included, as their sensitivity is low (especially during flu season) and false positives are common during low activity seasons.
* Laboratory-confirmed influenza through antibody assay as part of the primary outcome will not be included, as this is a less sensitive test than PCR and viral culture.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy subjects vaccinated with an influenza vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of laboratory-confirmed influenza [Polymerase Chain Reaction (PCR) or viral culture].

SECONDARY OUTCOMES:
Incidence of laboratory-confirmed influenza through antibody assay (a less sensitive test than PCR or viral culture), alone or combined with PCR, and/or viral culture.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline